CLINICAL TRIAL: NCT02037581
Title: Integrated Care in Early Psychosis (ICEP Study): a 12-month Quasi Experimental Study With Historic Control Group
Brief Title: Integrated Care Including Assertive Community Treatment in Early Psychosis
Acronym: ICEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Martin Lambert, Professor, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 01KQ1002B
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: integrated care; hometreatment; assertive community treatment (ACT); psychosis; schizophrenia; bipolar disorder; first episode
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early detection and Integrated Care (Experimental): The intervention condition consisted of measures to improve early detection and treatment quality (Integrated Care).
  1. Interventions for the improvement of early detection. The measures for improved early detection aiming at reducing the duration of untreated psychosis included 4-year measures to improve mental health literacy, reduce stigma and improve service utilization.
  2. Measures to improve treatment quality should be achieved through extending the Hamburg model to a cross-age and interdisciplinary Integrated Care model for adolescent and young adult patients with psychotic disorders aged 12-29 years.
  Interventions: Behavioral: Early detection and Integrated Care
- Standard Care (Other): Historical control group with standard care parallelized regarding age, diagnosis and illness stage, which was treated in the period before the implementation of the intervention conditions. The control group consisted of n=105 patients with early psychosis between the ages of 12 and 29, who had been treated between January 2005 and December 2008. The central differences in comparison with the intervention conditions lie in the lack of measures for the improvement of early detection, the absence of the TACT team, as well as the regular referral to an established psychiatrist with in most cases regular contact frequency.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Early detection and Integrated Care — Patients receive integrated care including therapeutic Assertive Community Treatment (TACT)
  Arms: Early detection and Integrated Care
Behavioral: Standard Care — Standard care as being offered by private psychiatrists
  Arms: Standard Care

SUMMARY:
Improvement of clinical long-term outcome through the implementation of early detection and intervention within a specialized network of integrated care (ACT and hometreatment) for adolescents and young adults with a first episode of psychosis between 12 and 29 years.

DETAILED DESCRIPTION:
The trial is carried out at the Psychosis Center of the Department of Psychiatry and Psychotherapy and the Department of Child and Adolescent Psychiatry at the University Medical Center Hamburg-Eppendorf (UKE), which has the responsibility to treat all Child, adolescent and adult patients within its catchment area of approximately 300.000 habitants.

The IC model was implemented into a network of the Psychosis Center of the University hospital (UKE), private psychiatrists and psychologists of the UKE catchment area and other outpatient facilities. As such, following health care structures are part of the model and could be used by each patients and its relatives according to need:

Specialized inpatient units with attached day-clinics for psychotic disorders; Acute inpatient units of both Departments; Specialized psychosis outpatient center with a variety of diagnosis-specific evidence-based individual- and group therapies, low-threshold offers to promote day structure (e.g., cooking, sport or art groups), an early detection and intervention service with a mobile early detection team with professionals from the child- and youth and adult psychiatry, possibility of peer-to-peer and relatives-to-relatives counseling, relative groups.

A multidisciplinary assertive community treatment (ACT) team, which was implemented according to guidelines of the Assertive Community Treatment Association and according to the Dartmouth Assertive Community Treatment Scale (DACTS). Compared to the traditional ACT model there are two important differences: (1) While traditional ACT models have a responsibility for patients with severe and persistent mental illness (SPMI) patients independent from the underlying diagnosis, the present model solely focus on patients with psychotic disorders; (2) The fidelity of the ACT team was further increased by composing a team of highly educated psychosis experts (i.e. consultant psychiatrists, psychiatrists, psychologists, nurses, social worker). Members of the ACT team received diagnosis-specific training in pharmacotherapy, cognitive behavioral (CBT), dynamic, and/or family psychotherapy.

A specialized day-clinic for first-episode psychosis patients in the age range of 15-29 years managed by the child- and youth and adult psychiatry; A working support outpatient center with outpatient and day-clinic treatment facilities; 20 private psychiatrists participate in the treatment network of the IC model (their duties and responsibilities are described below).

Further participants of the network are: a psychiatric nursing service, a specialized housing support service and a specialized psychosis living unit.

Within this network, the main responsibility for the individual patient and his relatives is generally allocated according to need and preferences to two specific members of the ACT team, of which one has to be a psychiatrist responsible for pharmacotherapy. However, when pharmacotherapy is stable and adherence assured, private psychiatrists are allowed to take over this responsibility. In this case, the specific IC contract with the private psychiatrists includes several quality assurance guidelines.

Briefly, the staff/client caseload ratio of a single full time employed ACT team member is 1:25. In any case, the first responsibility of the network is a broad assessment of the psychotic disorder, comorbid psychiatric and somatic disorders, traumatic events, previous service engagement and medication adherence, social problems, etc. Thereby, a need-adapted treatment plan will be developed together with the patient, relatives and other caregivers. If the patient starts IC during inpatient, transition from in- to outpatient care will be organized. Participant, relatives and other caregiver re-ceive two telephone numbers: one of the ACT therapists for all contacts within office hours (Monday to Friday from 8 am to 6 pm) and a 24 hours crisis number for all emergencies or questions outside office hours. The primary ACT/private psychiatrists subteam is responsible for high-frequent face-to-face treatment contacts fostering continuity of care, coordinating treatment and social support (case management), promoting and ensuring service engagement and medication adherence, and offering intensive need-adapted individual psychotherapy at the earliest possible time point. Crisis intervention is offered at any time and is always conducted by two ACT members of which one is the primary ACT therapist. Access to other need-adapted and diagnosis-specific evidence-based interventions is organized within the specialized psychosis outpatient center or the work support center, e.g. psychoeducation groups, social skills training, meta-cognitive training, bipolar psychotherapy groups, etc. Further, all low-threshold interventions in the outpatient center could be used at any time. Thereby day-clinic equivalent program could be organized while being in outpatient status. As many of these patients are at risk for service disengagement and medication non-adherence, a strict 'no-drop-out' policy is implemented including all admissions out of the catchment area.

Primary Outcome:

Rate of psychofunctional remission after 12 months of treatment in integrated care (ACT and hometreatment) versus standard care (SC, historic control group) for the treatment of adolescents and young adults with early psychosis (12-29 years)

Rationale:

The primary Outcome measure ist the number of patients with psychofunctional remission over at least 6 months(t2 - t1). Definition of symptomatic remission is according to the standardized remission criteria(siehe Andreasen et al. 2005). Functional remission is assessed as GAF ≥ 60. Psychofunctional remission is given, if both criteria are fulfilled through 6 months.

Secondary Outcomes:

Investigation of the effects of integrated care compared with standard care on:

A. Improvement of psychopathology, daily function and quality of life, B. Improevemnt of service engagement, compliance and satisfaction with care, C. Increase of Quality Adusted Life Years (QALY's) through 12 months of treatment.

D. Duration of untreated psychosis (DUP) and pathway of care

ELIGIBILITY:
Inclusion Criteria:

male/female, age 12-29, adequate knowledge of German language

1. Early psychosis critria according to Lewis, Tarrier, & Haddock, 2002 fullfilled: first or second hospitalisation for psychosis during the past 2 years, duration of illness (psychosis)≤2 years
2. Diagnosis chriteria according to DSM-IV TR fullfilled for schizophrenia(295.xx including all subtypes), schizophreniform psychosis(295.40), schizoaffektive disorder(295.70), delusional disorder (297.1), brief psychotic episode 298.8), psychotic disorder (298.9), bipolar I disorder (including 296.44, 296.54 and 296.64) and major depression with psychotic symptoms (296.24 and 296.34).

Exclusion Criteria:

One of the following diagnoses according to DSM-IV TR:

Alkcohol- or substance induced psychosis (z.B. 291.3, 291.5, 292.xx: -.11 or -.12); Psychosis according to somatic disorder(z.B. 293.0, 290.12, 290.20, 290.42, 293.89); pregnancy.

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Remission of psychosocial functioning | 12 months
  The primary outcome is the rate (yes / no in %) of patients with combined psycho-functional remission at 12 months study endpoint in the intervention (IC) versus the control condition (CC). The primary objective criterion was regarded as met when the following conditions were fulfilled:
  1. Symptomatic remission according to the criterion by Andreasen et al. [75]. In the ACCESS III study the criterion was regarded as fulfilled when a symptomatic remission was present at T2 (6 months) and T3 (12 months) and there had been no worsening of symptoms on one of the items in between.
  2. Functional remission pursuant to the criterion by Albert et al. [76]. In the ACCESS III study the criterion was regarded as fulfilled when a functional remission was present at T2 (6 months) and T3 (12 months) and there had been no worsening of functioning in between.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lambert, Prof., Study Director — UHH Hamburg-Eppendorf; Anne Karow, Prof., Study Chair — UHH Hamburg-Eppendorf
Locations (1):
- UHH Hamburg Eppendorf, Hamburg, Germany